CLINICAL TRIAL: NCT04629677
Title: Prospective Evaluation of Portal Vein (PV) Stenting in Patients With PV Stenosis and Gastrointestinal Malignancies
Brief Title: Evaluation of Portal Vein Stenting in Patients With Portal Vein Stenosis and Gastrointestinal Cancers
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PA18-0712; NCI-2020-07171 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA18-0712 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Malignant Digestive System Neoplasm
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A (questionnaire, medical record review): Patients complete a QoL questionnaire at 2-4 weeks and then 6-8 weeks after portal vein stenting procedure. Patients' medical records are also reviewed.
  Interventions: Other: Electronic Health Record Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Cohort B (medical record review): Patients' medical records are reviewed retrospectively.
  Interventions: Other: Electronic Health Record Review

INTERVENTIONS:
Other: Electronic Health Record Review — Review of medical records
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
  Groups: Cohort A (questionnaire, medical record review)
Other: Questionnaire Administration — Complete questionnaires
  Groups: Cohort A (questionnaire, medical record review)

SUMMARY:
This study collects information about the safety and effect of portal vein stenting in gastrointestinal cancer patients with portal vein stenosis. This study may help researchers learn how long the portal vein stays open and free from blockage and the effects of portal vein stenting on patients' overall well-being.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and efficacy of portal vein stenting in patients with portal vein (PV) stenosis and gastrointestinal malignancies, including quality of life measurements.

SECONDARY OBJECTIVES:

I. Stent patency and duration of clinical success related to the intervention. II. Compare the efficacy of portal vein stenting on liver volumes, nutritional status, and laboratory values relative to patients with portal vein stenosis/thrombosis who do not undergo portal vein stenting.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT A: Patients complete a quality of life (QoL) questionnaire at 2-4 weeks and then 6-8 weeks after portal vein stenting procedure. Patients' medical records are also reviewed.

COHORT B: Patients' medical records are reviewed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* COHORT A: All patients will undergo initial staging and treatment as per the institution standard of care. Patients will be considered eligible for porto-mesenteric venous stenting (PVS) if:

  * There is > 75% porto-mesenteric venous stenosis in either main portal vein (PV), left PV, right PV, or the superior mesenteric vein (SMV), even in absence of symptoms of portal hypertension
  * Patients presented with any degree of vascular narrowing of said vessels and symptomatic portal hypertension including variceal bleeding, refractory ascites, abdominal pain, intestinal edema, or diarrhea after exclusion of tumor-related causes as direct tumor invasion or peritoneal dissemination
* COHORT B: Patients who have thrombosis/stenosis of the main portal vein but who did not undergo stenting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastrointestinal cancer patients with portal vein stenosis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Patency rate (Cohort A) | Up to 8 weeks after stent placement
  Defined by successful stent placement and described as N (%) of patients with corresponding exact 95% confidence interval.
Transfusion rate (Cohort A) | Up to 8 weeks after stent placement
  N (%) of patients receiving transfusion with corresponding exact 95% confidence interval. Instances of multiple transfusions per patient will also be described.
Rate of paracenteses for ascites (Cohort A) | Up to 8 weeks after stent placement
  N (%) of patients receiving paracenteses with corresponding exact 95% confidence interval. Instances of multiple paracenteses per patient will also be described.
Duration of clinical success (Cohort A) | Up to 8 weeks after stent placement
  Mean, median, standard deviation, and minimum/maximum values will be described.
Change in nutritional status (Cohort A) | Baseline up to 30 days post procedure
  Based on albumin, pre-albumin, weight, body fat, and body surface area (BSA). Methods such as repeated measures analysis of variance (ANOVA) with post-hoc Tukey test and generalized estimating equations (GEE) will be used to assess pre- and post- differences.
Change in bleeding risk (Cohort A) | Baseline up to 30 days post procedure
  Based on platelet count and coagulation factors. Methods such as repeated measures ANOVA with post-hoc Tukey test and GEE will be used to assess pre- and post- differences.
Change in liver function (Cohort A) | Baseline up to 30 days post procedure
  Methods such as repeated measures ANOVA with post-hoc Tukey test and GEE will be used to assess pre- and post- differences.
Change in liver volume (Cohort A) | Baseline up to 30 days post procedure
  Methods such as repeated measures ANOVA with post-hoc Tukey test and GEE will be used to assess pre- and post- differences.
Change in quality of life (QoL) (Cohort A) | Baseline up to 30 days post procedure
  Will be assessed based on National Comprehensive Cancer Network - Hepatibiliary Symptom Index Questionnaire - 18 item. Methods such as repeated measures ANOVA with post-hoc Tukey test and GEE will be used to assess pre- and post- differences. For QoL will also present effect size, defined as the magnitude of the differences in relation to the standard deviation of the scores, which will be reflective of the strength of the effect of portal stenting on QoL.
Number of transfusions (Cohort A and B) | Up to 8 weeks post procedure
  Methods such as paired t-tests, conditional logistic regression, and generalized linear modeling will be used to compare differences by cohort.
Number of paracentesis for ascites (Cohort A and B) | Up to 8 weeks post procedure
  Methods such as paired t-tests, conditional logistic regression, and generalized linear modeling will be used to compare differences by cohort.
Liver volume (Cohort A and B) | Up to 8 weeks post procedure
  Methods such as paired t-tests, conditional logistic regression, and generalized linear modeling will be used to compare differences by cohort.
Liver function (Cohort A and B) | Up to 8 weeks post procedure
  Methods such as paired t-tests, conditional logistic regression, and generalized linear modeling will be used to compare differences by cohort.
Nutritional status (Cohort A and B) | Up to 8 weeks post procedure
  Based on albumin, pre-albumin, weight, body fat, and BSA. Methods such as paired t-tests, conditional logistic regression, and generalized linear modeling will be used to compare differences by cohort.
Bleeding risk (Cohort A and B) | Up to 8 weeks post procedure
  Based on platelet count and coagulation factors. Methods such as paired t-tests, conditional logistic regression, and generalized linear modeling will be used to compare differences by cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Kuban, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org